CLINICAL TRIAL: NCT04620148
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Proof-of-Concept, Phase 2a Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous TAK-242 in Subjects With Acute Alcoholic Hepatitis Causing Decompensation of Alcohol-related Cirrhosis and Acute-on-Chronic Liver Failure
Brief Title: TAK-242 in Patients With Acute Alcoholic Hepatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akaza Bioscience Ltd (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-242-2001
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — ethyl 6-(N-(2-chloro-4-fluorophenyl)sulfamoyl)cyclohex-1-ene-1-carboxylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-242 (Experimental): Patients will be administered TAK-242 as a continuous IV infusion with standard care starting with a loading dose of 0.9 mg/kg administered over 30 minutes, followed by a continuous, constant rate infusion of 1.8 mg/kg/day for 7 days
  Interventions: Drug: TAK-242
- Placebo (Placebo Comparator): Patients will be administered placebo as a continuous IV infusion with standard care starting with a loading dose of 0.9 mg/kg administered over 30 minutes, followed by a continuous, constant rate infusion of 1.8 mg/kg/day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-242 — TAK-242 concentrate solution 80 mg/mL for dilution and infusion
  Arms: TAK-242
Drug: Placebo — Matching placebo concentrate solution
  Arms: Placebo

SUMMARY:
A phase 2a double-blind, randomized, placebo-controlled, multicenter, proof-of-concept study to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of TAK-242 in subjects with acute decompensation of alcohol-related cirrhosis due to alcoholic hepatitis resulting in acute-on-chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* History of alcohol-related cirrhosis who continue to drink heavily
* History of an acute decompensating event with a clinical and/or liver biopsy diagnosis of alcoholic hepatitis
* Grade 1 or 2 ACLF using the CLIF-C OF score; OR bilirubin criteria OR criteria of acute kidney injury Stage 1b or 2 after initial supportive treatment with fluids, albumin, or terlipressin; AND CLIF-C ACLF score is >35 and <64
* History of alcohol-related cirrhosis based on clinical, radiological, and/or histological evidence

Exclusion Criteria:

* Received certain previous therapies (any investigational drug within 30 days of randomization, corticosteroids for alcohol-induced liver failure within 4 weeks of randomization, or received TAK-242 in any previous study)
* History of liver cirrhosis from other chronic diseases; liver failure from other causes
* History of liver transplantation, post-operative decompensation after partial hepatectomy, acute or subacute liver failure without underlying cirrhosis
* Any untreated infections including gram-positive infections, or active or latent atuberculosis, sepsis or septic shock, or coinfection with hepatitis B virus, hepatitis C virus, hepatitis E virus, or HIV
* Chronic or pre-existing kidney failure, uncontrolled medical disorder that might confound study results or compromise subject safety, oxygen saturation <90%, or requires mechanical ventilation.
* Uncorrected anemia, methemoglobinemia, disseminated intravascular coagulation, significant or uncontrolled bleeding, atypical laboratory screening tests.
* Uncontrolled seizures, Grade 3 or 4 hepatic encephalopathy, Creutzfeldt-Jakob disease, glucose-6-phosphate dehydrogenase deficiency.
* Active extrahepatic malignancy or survival prognosis of <6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in CLIF-C ACLF score from baseline to Day 8 | Baseline to Day 8

SECONDARY OUTCOMES:
Percentage of subjects who experience at least 1 markedly abnormal treatment-emergent AE or SAE | To Day 28
  The percentage of subjects who experience at least 1 treatment-emergent AE or SAE that meets the Sponsor's markedly abnormal criteria
Percentage of subjects who experience at least 1 treatment-emergent clinical laboratory test result or abnormal ECG that meets the Sponsor's markedly abnormal criteria | To Day 28
  The percentage of subjects who experience at least 1 treatment-emergent clinical laboratory test result or abnormal ECG that meets the Sponsor's markedly abnormal criteria
Percentage of subjects who discontinue study drug due to an AE | To Day 28
Change in naturally log-transformed key biomarkers | Baseline to day 8
  Change in naturally log-transformed key biomarkers (TB, IL-8, high sensitivity CRP [hs-CRP], and urinary NGAL)
Survival at Day 28 after initiation of TAK-242 therapy versus placebo | Baseline to Day 28

IPD SHARING:
Plan to Share IPD: No